CLINICAL TRIAL: NCT01767129
Title: A Phase 2a, Double-blind, Randomized, Placebo-controlled, Crossover Study to Evaluate the Safety and Efficacy of AVP-923 (Dextromethorphan/Quinidine) in the Treatment of Levodopa-induced Dyskinesia in Parkinson's Disease Patients.
Brief Title: Safety and Efficacy of AVP-923 in the Treatment of Levodopa-induced Dyskinesia in Parkinson's Disease Patients
Acronym: LID in PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-AVR-133
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Results first posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Dyskinesia; Parkinson's Disease
Keywords: levodopa; dyskinesia; parkinson's disease; AVP-923; dextromethorphan; quinidine
MeSH Terms: conditions — Dyskinesias; Parkinson Disease | interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AVP-923-45 (Experimental): AVP-923-45 twice daily for 14 days
  Interventions: Drug: AVP-923-45
- Placebo (Placebo Comparator): Placebo twice a day for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVP-923-45 — One capsule twice daily for 14 days
  Other Names: dextromethorphan/quinidine
  Arms: AVP-923-45
Drug: Placebo — One capsule twice daily for 14 days
  Arms: Placebo

SUMMARY:
To evaluate the efficacy, safety, and tolerability of AVP-923 capsules containing 45 mg dextromethorphan and 10 mg quinidine (AVP-923-45) compared to placebo for the treatment of levodopa-induced dyskinesia (LID) in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Proof-of-concept phase 2a, double-blind, randomized, placebo-controlled, crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 30 to 80 years of age, inclusive.
* Diagnosis of idiopathic PD meeting the United Kingdom Parkinson's disease Society Brain Bank criteria.
* Levodopa-induced dyskinesia present greater than 25% of the day as per MDS-UPDRS.
* Dyskinesia of at least moderate severity as per MDS-UPDRS
* Amantadine and Monoamine Oxidase (MAO) inhibitors must be discontinued at least three weeks prior to randomization.
* Subjects currently receiving anti-parkinsonian medications, including all Levodopa preparations are eligible provided they have been on a stable dose of these medications for at least 1 month prior to randomization.
* Concomitant use of antidepressants such as selective serotonin reuptake inhibitors are allowed, provided the dose has been stable for at least 1 month prior to randomization.

Exclusion Criteria:

* Subject had a prior surgery for PD except Deep Brain Stimulation (Deep Brain Stimulation must not have been performed within one year of screening)
* Hoehn and Yahr score of 5 when "off".
* Subject with Cognitive impairment and/or history of psychiatric manifestations or active hallucinations.
* Subjects with any history of complete heart block, QTc prolongation, or torsades de pointes.
* Subjects with any family history of congenital QT interval prolongation syndrome.
* Subjects with history of postural syncope, or any history of unexplained syncope within the last 12 months.
* Subjects with a history of substance and/or alcohol abuse within the past 2 years.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2015-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Chicago, Illinois
  - Portland, Oregon
- Toronto, Ontario, Canada

REFERENCES:
- [Result] Fox SH, Metman LV, Nutt JG, Brodsky M, Factor SA, Lang AE, Pope LE, Knowles N, Siffert J. Trial of dextromethorphan/quinidine to treat levodopa-induced dyskinesia in Parkinson's disease. Mov Disord. 2017 Jun;32(6):893-903. doi: 10.1002/mds.26976. Epub 2017 Mar 30. PMID 28370447
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28370447/

RESULTS

PARTICIPANT FLOW:
Groups:
- AVP-923-45; Placebo: In Treatment Period 1, participants received one AVP-923-45 (45 milligrams [mg] dextromethorphan hydrobromide [DM]/10 mg quinidine sulfate [Q]) capsule once daily in the morning for 3 days, then twice daily, approximately 12 hours apart, for 11 days. In Treatment Period 2, participants received one placebo capsule once daily in the morning for 3 days, then twice daily, approximately 12 hours apart, for 11 days. The two treatment periods were separated by a 14-day washout period.
- Placebo; AVP-923-45: In Treatment Period 1, participants received one placebo capsule once daily in the morning for 3 days, then twice daily, approximately 12 hours apart, for 11 days. In Treatment Period 2, participants received one AVP-923-45 capsule once daily in the morning for 3 days, then twice daily, approximately 12 hours apart, for 11 days. The two treatment periods were separated by a 14-day washout period.
Period: Treatment Period 1 (14 Days)
Arm/Group | AVP-923-45; Placebo | Placebo; AVP-923-45
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Treatment Period 2 (14 Days)
Arm/Group | AVP-923-45; Placebo | Placebo; AVP-923-45
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were randomized to receive AVP-923-45 (45 milligrams [mg] dextromethorphan hydrobromide [DM]/10 mg quinidine sulfate [Q]) and placebo in one of two treatment sequences: AVP-923-45 in Treatment Period 1, placebo in Treatment Period 2; or placebo in Treatment Period 1, AVP-923-45 in Treatment Period 2. The two treatment periods were separated by a 14-day washout period. In both treatment periods, participants received either one AVP-923-45 capsule or one placebo capsule once daily in the morning for 3 days, then twice daily, approximately 12 hours apart, for 11 days.
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13
  Indian Sub-Continent | 1

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Dyskinesia Severity Area Under the Curve (AUC) Score As Assessed By Modified Movement Disorder Society-Unified Dyskinesia Rating Scale (MDS-UDysRS) Part 3
Description: The MDS-UDysRS was developed to evaluate involuntary movements often associated with treated Parkinson's disease (PD). Levodopa-Induced Dyskinesia severity was assessed via video analysis by unbiased blinded central raters, and was calculated using the Intensity Scale from Part 3 of the MDS-UDysRS. The Intensity Scale was made up of seven body parts: face, neck, right arm/shoulder, left arm/shoulder, trunk, right leg/hip, and left leg/hip. Each body part was scored on a variety of disability items (communication, drinking, and ambulation [walking]) on a scale of 0 (normal) to 4 (incapacitating dyskinesia) with a maximum total score of 28. For each body part, the highest disability score was summed to calculate the intensity score. A score of '0' was assigned to questions associated with the dressing task which were not performed due to the placement of the treatment infusion (IV) line. A higher score indicated more severe symptoms.
Time Frame: Over the 2-hour levodopa infusion period on the last day of each treatment period (Day 14 and Day 42)
Population: Efficacy Evaluable (EE) Population: all randomized participants who completed the study
Measure: Least Squares Mean (Standard Error); unit: (Score on a scale)*hour
Groups:
- AVP-923-45: Participants received one AVP-923-45 capsule (45 milligrams [mg] dextromethorphan hydrobromide [DM]/10 mg quinidine sulfate [Q]) once daily in the morning for 3 days, then twice daily, approximately 12 hours apart, for 11 days in either Treatment Period 1 or Treatment Period 2. The two treatment periods were separated by a 14-day washout period.
- Placebo: Participants received one placebo capsule once daily in the morning for 3 days, then twice daily, approximately 12 hours apart, for 11 days in either Treatment Period 1 or Treatment Period 2. The two treatment periods were separated by a 14-day washout period.
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
(Score on a scale)*hour | 966.0 (42.22) | 1049.4 (42.22)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Test type: Superiority; p = 0.1907, ANOVA; The standard analysis of variance (ANOVA) model for a 2-period crossover trial was used. Factors in the model were participant, treatment, and period; Mean Difference (Final Values) = -83.4, 95% CI 2-sided [-215.02 to 48.23] — The least squares (LS) mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

2. Secondary Outcome: Least Squares Mean Disability Area Under the Curve (AUC) Score As Assessed By Modified Movement Disorder Society-Unified Dyskinesia Rating Scale (MDS-UDysRS) Part 4
Description: The MDS-UDysRS was developed to evaluate involuntary movements often associated with treated PD. Part 4 of the MDS-UDysRS objectively measures the disability associated with levodopa-induced dyskinesia. Disability was assessed via video analysis by unbiased blinded central raters. Disability was evaluated for communication, drinking from a cup, and ambulation items. Each item was rated from 0 (no dyskinesia) to 4 (most severe disability), with a sum range of 0 to 12. A score of '0' was assigned to questions associated with the dressing task because it was not performed due to placement of the IV line. A higher score indicated more severe symptoms.
Time Frame: Over the 2-hour levodopa infusion period on the last day of each treatment period (Day 14 and Day 42)
Population: EE Population
Measure: Least Squares Mean (Standard Error); unit: (Score on a scale)*hour
Groups:
- AVP-923-45: Participants received one AVP-923-45 capsule once daily in the morning for 3 days, then twice daily, approximately 12 hours apart, for 11 days in either Treatment Period 1 or Treatment Period 2. The two treatment periods were separated by a 14-day washout period.
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
(Score on a scale)*hour | 409.4 (14.87) | 428.3 (14.87)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Test type: Superiority; p = 0.3880, ANOVA; The standard ANOVA model for a 2-period crossover trial was used. Factors in the model were participant, treatment, and period; Median Difference (Final Values) = -18.9, 95% CI 2-sided [-65.28 to 27.42] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

3. Secondary Outcome: Least Squares Mean Motor Movement Area Under the Curve Score As Assessed by Modified Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part III
Description: The Modified MDS-UPDRS (4 parts) was used to assess the severity of parkinsonian disability. Part III of the MDS-UPDRS was used as an objective measure of the severity of parkinsonian disability per motor examination with focus on the treated side tremor and motor fluctuations. The motor examination were videotaped using a standardized protocol for review by an expert central rater blinded to the treatment schedule. A total of 11 items were scored as follows: 0 (normal), 1 (slight), 2 (mild), 3 (moderate), 4 (severe), with a maximum total score of 44. For each part, a higher score indicated more severe symptoms. Due to placement of the IV line, a score of '0' was assigned to rigidity questions.
Time Frame: Over the 2-hour levodopa infusion period on the last day of each treatment period (Day 14 and Day 42)
Population: EE Population
Measure: Least Squares Mean (Standard Error); unit: (Score on a scale)*hour
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
(Score on a scale)*hour | 6568.9 (383.26) | 6397.0 (383.26)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Test type: Superiority; p = 0.7574, ANOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 171.9, 95% CI 2-sided [-1022.79 to 1366.64] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

4. Secondary Outcome: Least Squares Mean Timed Finger Tapping Area Under the Curve (AUC) Score
Description: Timed finger tapping test was used to quantify the upper extremity impairment in participants with idiopathic PD. Timed finger tapping was assessed using the Objective Parkinson's Disease Measurement (OPDM) System. Participants were instructed to tap for 60 seconds while speed and accuracy were assessed across 4 tests; right and left two finger test (m,n keystrokes) and one finger test (p,q keystrokes). The mean peak finger tapping score was calculated using the individual peak values. A higher score signifies improvement (faster typing, more accuracy), while a lower score signifies increased symptom severity.
Time Frame: Over the 2-hour levodopa infusion period on the last day of each treatment period (Day 14 and Day 42)
Population: EE Population
Measure: Least Squares Mean (Standard Error); unit: (Score on a scale)*hour
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
(Score on a scale)*hour | 820.9 (40.80) | 772.1 (40.80)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Test type: Superiority; p = 0.4203, ANOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 48.8, 95% CI 2-sided [-80.63 to 178.30] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

5. Secondary Outcome: Change From Baseline in MDS-UPDRS Scores for Part I, II, and IV
Description: The MDS-UPDRS was used to assess the status of PD. Parts I and II (completed by the participant) and Part IV (completed by a rater) of the MDS-UPDRS provided a subjective measure of parkinsonian disability. Part I measured non-motor experiences of daily living, Part II measured motor experiences of daily living, and Part IV measures motor complications associated with PD. Each part was comprised of a series of questions, and each question was scored from 0 (normal) to 4 (severe). Part I and Part II were each comprised of 13 items; the total score ranges from 0 (normal) to 52 (severe). Part III was comprised of 33 items; the total score ranges from 0 (normal) to 132 (severe). Part IV was comprised of 6 items; the total score ranged from 0 (normal) to 24 (severe). For each part, a higher score indicated more severe symptoms. Post-Baseline was Visit 2 (Day 14) or Visit 4 (Day 42). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1); Post-Baseline (Day 14 or 42)
Population: EE Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
score on a scale
  Part I | -1.2 (0.43) | -0.1 (0.43)
  Part II | -0.0 (0.92) | -0.2 (0.92)
  Part IV | -2.9 (0.84) | -0.5 (0.84)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Part I; Test type: Superiority; p = 0.1067, ANOVA; Change from Day 1 values were compared using ANOVA for a 2-period crossover trial. Factors in the model were participant, treatment, and period; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.41 to 0.27] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 2: Comparison: AVP-923-45 vs Placebo; Part II; Test type: Superiority; p = 0.8650, ANOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-2.64 to 3.09] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 3: Comparison: AVP-923-45 vs Placebo; Part IV; Test type: Superiority; p = 0.0745, ANOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-4.94 to 0.27] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

6. Secondary Outcome: Change From Baseline in MDS-UDysRS Scores for Part 1 and 2
Description: The MDS-UDysRS was developed to evaluate involuntary movements often associated with treated PD. Part 1 (On-Dyskinesia ['jerking or twisting movements that occur when your medicine is working']) and Part 2 (Off-Dyskinesia ["spasms or cramps that can be painful and occur when your PD medications are not taken or are not working]) of the MDS-UDysRS were assessed by a blinded rater. Parts 1B and 2B (participant questionnaires) were completed at home by the participant. Part 1 comprised of 11 items, and Part 2 comprised of 4 items. All items were assigned a score of: 0, normal; 1, slight; 2, mild; 3, moderate; 4, severe. The total score for Parts 1 and 2 ranged from 0 to 44 and from 0 to 16, respectively. Higher scores indicate increased symptom severity. Post-Baseline was Visit 2 (Day 14) or Visit 4 (Day 42). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1); Post-Baseline (Day 14 or 42)
Population: EE Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
score on a scale
  Part 1 | -3.9 (1.34) | 0.00 (1.34)
  Part 2 | -0.7 (0.77) | 0.6 (0.77)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Part 1; Test type: Superiority; p = 0.0625, ANOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-8.10 to 0.24] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 2: Comparison: AVP-923-45 vs Placebo; Part 2; Test type: Superiority; p = 0.2474, ANOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.74 to 1.07] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

7. Secondary Outcome: Change From Baseline in PD Motor Diary Ratings Of Duration Of "On-time Without Bothersome Dyskinesia"
Description: The PD motor diary is a home diary used to assess functional status in participants with PD with motor fluctuations and dyskinesia. Participants were instructed to complete the PD motor diary at home for a minimum of 3 consecutive days within the 7 days prior to Visits 2 and 4 (Days 14 and 42). Baseline is Visit 1 (Day 1) or Visit 3 (Day 29); Post-Baseline is Visit 2 (Day 14) or Visit 4 (Day 42). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Post-Baseline (Days 14 and 42)
Population: EE Population
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
hours | 0.5 (1.01) | 0.5 (0.93)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Test type: Superiority; p = 0.9764, ANOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-3.10 to 3.01] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

8. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire-39 (PDQ-39) Domain Scores at the End of Each Treatment Period
Description: The PDQ-39 was a self-reported questionnaire consisting of 39 questions assessing Parkinson's disease-specific health quality of life covering 8 aspects of quality of life: mobility; activities of daily living; emotional wellbeing; stigma; social support; cognitive impairment (cognitions); communication; bodily discomfort. Each item was scored on 5-point scale: 0 = Never (better in outcome), 1 = Occasionally, 2 = Sometimes, 3 = Often, 4 = Always (worse in outcome). Total scores ranged between 0 to 156. Higher scores indicated poor quality of life. Baseline was Visit 1 (Day 1) or Visit 3 (Day 29); Post-Baseline was Visit 2 (Day 14) or Visit 4 (Day 42). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Post-Baseline (Day 14 or 42)
Population: EE Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
score on a scale
  Mobility | 0.2 (2.45) | 2.0 (2.69)
  Activities of Daily Living | -4.6 (2.14) | 3.9 (2.14)
  Emotional Well Being | -4.5 (2.90) | 2.9 (2.90)
  Stigma | -3.7 (4.10) | 0.3 (4.10)
  Social support | -6.0 (3.60) | 3.8 (3.60)
  Cognitive impairment (Cognitions) | -4.1 (3.64) | 0.2 (3.64)
  Communication | -3.7 (2.43) | 2.4 (2.43)
  Bodily discomfort | -7.4 (4.60) | -2.2 (4.60)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Mobility; Test type: Superiority; p = 0.6359, ANOVA; Change from Baseline values were compared using ANOVA for a 2-period crossover trial. Factors in the model were participant, treatment, and period; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-9.94 to 6.36] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 2: Comparison: AVP-923-45 vs Placebo; Activities of Daily Living; Test type: Superiority; p = 0.0167, ANOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-15.20 to -1.87] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 3: Comparison: AVP-923-45 vs Placebo; Emotional Well Being; Test type: Superiority; p = 0.0959, ANOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-16.54 to 1.56] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 4: Comparison: AVP-923-45 vs Placebo; Stigma; Test type: Superiority; p = 0.5108, ANOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-16.72 to 8.83] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 5: Comparison: AVP-923-45 vs Placebo; Social support; Test type: Superiority; p = 0.0806, ANOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -9.8, 95% CI 2-sided [-21.06 to 1.42] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 6: Comparison: AVP-923-45 vs Placebo; Cognitive impairment (Cognitions); Test type: Superiority; p = 0.4205, ANOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-15.66 to 7.03] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 7: Comparison: AVP-923-45 vs Placebo; Communication; Test type: Superiority; p = 0.1065, ANOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-13.63 to 1.53] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 8: Comparison: AVP-923-45 vs Placebo; Bodily discomfort; Test type: Superiority; p = 0.4456, ANOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -5.2, 95% CI 2-sided [-19.51 to 9.19] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

9. Secondary Outcome: Change From Baseline in PDQ-39 Single Index (PDQ-39-SI) Scores at the End of Each Treatment Period
Description: The PDQ-39 was the most widely used PD-specific measure of health status. It consists of 39 questions, covering 8 aspects of quality of life: mobility; activities of daily living; emotional wellbeing; stigma; social support; cognitive impairment (cognitions); communication; bodily discomfort. The instrument was developed on the basis of interviews with people diagnosed with PD. The PDQ-39-SI) score was calculated as the weighted addition of scores on all 8 dimensions of the PDQ-39. The total score ranged from 0 (no disease impact) to 100 (severe disease impact). Baseline was Visit 1 (Day 1) or Visit 3 (Day 29); Post-Baseline was Visit 2 (Day 14) or Visit 4 (Day 42). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Post-Baseline (Day 14 or 42)
Population: EE Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
score on a scale | -4.2 (1.60) | 2.2 (1.76)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Test type: Superiority; p = 0.0233, ANOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-11.72 to -1.07] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

10. Secondary Outcome: Change From Screening in the Montreal Cognitive Assessment (MoCA) Calculated Score at the End of Each Treatment Period
Description: The MoCA was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total score is calculated by summing the items from each domain. Total scores can range from 0 to 30; lower scores indicate cognitive dysfunction. A final total score of 26 and above is considered normal. Change from Screening was calculated as the post-Screening value minus the Screening value.
Time Frame: Screening (Day -28); End of each treatment period (Days 14 or 42)
Population: EE Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
score on a scale | 0.1 (0.27) | 0.6 (0.27)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Test type: Superiority; p = 0.1930, ANOVA; Change from Screening values were compared using ANOVA for a 2-period crossover trial. Factors in the model were participant, treatment, and period; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.39 to 0.31] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

11. Secondary Outcome: Change From Baseline in the Dyskinesia and Other PD Symptoms Score As Assessed by Patient Global Impression of Change (PGIC)
Description: The PGIC was a 7-point scale used to assess treatment response as judged by the participant. The participant was asked to assess change in dyskinesia symptoms and change in overall PD symptoms (e.g., slowness, stiffness, balance) on a score range of 1, much improved; 2, improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, worse; 7, much worse. The average PGIC score was calculated at each visit by treatment group. Baseline is Visit 1 (Day 1) or Visit 3 (Day 29); Post-Baseline is Visit 2 (Day 14) or Visit 4 (Day 42). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Post-Baseline (Days 14 and 42)
Population: EE Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AVP-923-45 | Placebo
Number analyzed (Participants) | 13 | 13
score on a scale
  Dyskinesia | 2.7 (0.35) | 3.7 (0.35)
  Other PD symptoms | 4.2 (0.26) | 4.1 (0.26)
Statistical Analysis 1: Comparison: AVP-923-45 vs Placebo; Dyskinesia; Test type: Superiority; p = 0.0511, ANOVA; Change were compared using ANOVA for a 2-period crossover trial. Factors in the model were participant, treatment, and period; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.17 to 0.01] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean
Statistical Analysis 2: Comparison: AVP-923-45 vs Placebo; Other symptoms; Test type: Superiority; p = 0.7745, ANOVA; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.70 to 0.91] — The LS mean difference was calculated as the AVP-923-45 LS mean minus the placebo LS mean

ADVERSE EVENTS:
Time Frame: up to Day 42
Description: TEAEs, defined as events that began on or after the first dose of study drug up until 30 days after the last dose, are reported. TEAEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of study treatment.
Arm/Group | AVP-923-45 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 11/14 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AVP-923-45 (N=14) | Placebo (N=13)
Palpitations (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Freezing phenomenon (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Male sexual dysfunction (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other